CLINICAL TRIAL: NCT01197027
Title: Feasibility and Acceptability Study of an Individual-Level Behavioral Intervention for Individuals With Acute and Early HIV-Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HIV Prevention Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HPTN 062
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Acute HIV Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced counseling (Experimental): 5 intensive counseling sessions following acute HIV infection
  Interventions: Behavioral: Standard counseling
- Standard counseling (Active Comparator): Standard HIV counseling following acute HIV infection
  Interventions: Behavioral: Standard counseling

INTERVENTIONS:
Behavioral: Standard counseling — Standard HIV counseling

SUMMARY:
The purpose of this study is to evaluate the acceptability and feasibility of an enhanced, individual-level counseling intervention for individuals in the acute and early phase of HIV infection aimed at reducing risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Be enrolled in CHAVI 001 Note: The inclusion and exclusion criteria for CHAVI 001 are provided below. The criteria will not be reassessed prior to enrollment in HPTN 062.
* Inclusion Criteria from CHAVI 001

  * Men and women aged ≥ 18 years at the time of screening.
  * Able and willing to provide adequate information for locator purposes.
  * Hemoglobin > 10.0 g/dL.
  * Willing to receive HIV test results.
  * Not intending to relocate out of the area for the duration of study participation and does not have a job or other obligations that may require long absences from the area.
  * Has acute HIV infection. (See Section 2.3 for definition).

Exclusion Criteria:

* Any prior or current use of antiretroviral therapy (ART). This does not apply to individuals screening for Group 1A. ART use for the prevention of perinatal transmission may be waived after prior consultation with the protocol team.

  * Previous or current participation in a HIV vaccine study. HPTN 062 Version 3.0 Final 03 August 2010
  * Any condition that, in the opinion of the Investigator of Record, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-02; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Proportion of participants in the experimental arm who receive the first four intervention sessions between enrollment and week 2 visit | Week 2

SECONDARY OUTCOMES:
Number of self-reported unprotected sex acts | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Amy Corneli, PhD, Study Chair — FHI 360; Audrey Pettifor, PhD, Study Chair — FHI 360; Francis Martinson, Md, PhD, Principal Investigator — Kamuzu Central Hospital
Locations (1):
- Kamuzu Central Hospital, Lilongwe, Malawi

REFERENCES:
- [Derived] Pettifor A, Corneli A, Kamanga G, McKenna K, Rosenberg NE, Yu X, Ou SS, Massa C, Wiyo P, Lynn D, Tharaldson J, Golin C, Hoffman I; HPTN 062 Study Protocol Team. HPTN 062: A Pilot Randomized Controlled Trial Exploring the Effect of a Motivational-Interviewing Intervention on Sexual Behavior among Individuals with Acute HIV Infection in Lilongwe, Malawi. PLoS One. 2015 May 11;10(5):e0124452. doi: 10.1371/journal.pone.0124452. eCollection 2015. PMID 25962118